CLINICAL TRIAL: NCT00002253
Title: A Multicenter Placebo-Controlled Double Blind Study to Evaluate the Efficacy and Safety of Sandostatin ( SMS 201-995 ) in Patients With Acquired Immunodeficiency Related Diarrhea Who Were Either "Responders" or "Non-Responders" in a Prior Placebo-Controlled Double-Blind Sandostatin Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 102B; D204
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-08

CONDITIONS: Diarrhea; HIV Infections
Keywords: Octreotide; Diarrhea; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Diarrhea; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
The primary objective of this study is to determine the relapse rate in patients with AIDS-related diarrhea who were found to be "Responders" in a previous placebo-controlled, double-blind study of Sandostatin (Study #D203 - FDA 102A).

The secondary objectives include: 1) To evaluate clinical efficacy and safety of open-label Sandostatin in patients who were "Non-Responders" in Study #D203 - FDA 102A; 2) To evaluate the efficacy and safety of Sandostatin during prolonged open-label treatment in "Responders" from Study #D03 - FDA 102A.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Only patients who have completed the duration of Study D203, FDA 102A will be eligible for this study.
* Each of these patients must give written informed consent to participate in Study D204, FDA 102B as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - USC School of Medicine, Los Angeles, California
  - UCSD Med Ctr, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - San Mateo County Gen Hosp, San Mateo, California
  - Med Service, Miami, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Maine Med Ctr Med Clinics, Portland, Maine
  - Douglas Plesko, Boston, Massachusetts
  - Boston City Hosp, Boston, Massachusetts
  - Henry Ford Hosp, Detroit, Michigan
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Mount Sinai Med Ctr, New York, New York
  - SUNY Stony Brook / Health Sciences Ctr, Stony Brook, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Miriam Hosp / Family Healthcare Ctr at SSTAR, Providence, Rhode Island
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Wisconsin School of Medicine, Madison, Wisconsin